CLINICAL TRIAL: NCT04457037
Title: Treatment of Patients With Trophic Ulcers Using Autologous Adipose-derived Mesenchymal Stem Cells
Brief Title: Treatment of Patients With Trophic Ulcers Using Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(TrophicUlcer)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Trophic Ulcer
Keywords: Trophic Ulcer; Mesenchymal stem cells

STUDY DESIGN:
Intervention Model Description: Patients with trophic ulcers received standard treatment and mesenchymal stem cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC (Experimental): Patients with trophic ulcers received standard treatment and MSC
  Interventions: Biological: Autologous adipose-derived mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem cells — Autologous adipose-derived mesenchymal stem cells

SUMMARY:
Treatment of patients with trophic ulcers using injection of autologous adipose-derived mesenchymal stem cells around and inside the wound

DETAILED DESCRIPTION:
During the implementation of the project, it was planned to develop a method for the treatment of trophic ulcers using injection of autologous adipose-derived mesenchymal stem cells in the wound. The positive outlook for the effectiveness of MSCs is due to the following:

* the ability of MSCs to stimulate tissue regeneration
* positive results of preclinical studies of the method of treatment of trophic ulcers in animals (rats).

In study were included 18 patients (28 trophic ulcers treated). MSCs will be isolated from adipose tissue, cultured and then transplanted back to the wound. From 1 to 10 million MSCs in 4 ml were injected depending on the area of the wound. Follow up patients monitoring will occur at 1，2 and 3, 6, 12, 22 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Trophic Ulcers

Exclusion Criteria:

* diagnosed cancer
* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with tropic ulcers cured | 1 month
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  MSC injection related adverse events assessed by blood count and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor Volotovski, Dr, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Stanislav Tretyak, Prof, Study Director — Head of 2 Department of Surgical Diseases of BSMU
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No